CLINICAL TRIAL: NCT01095627
Title: Characterization of Aerosol Generation and Transport in the Human Lung of Subjects With Mild Intermittent Allergic Asthma Before and After Methacholine Challenge
Brief Title: Characterization of Aerosol Generation and Transport in the Human Lung
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fraunhofer-Institute of Toxicology and Experimental Medicine (Other)
Responsible Party: Prof. Dr. Norbert Krug, Fraunhofer-Institute of Toxicology and Experimental Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 10/04 AEROB
Record Dates: First submitted 2010-03-12; First posted 2010-03-30 (Estimated); Last update posted 2011-02-09 (Estimated); Status verified 2011-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Metacholine Challenge (Other): Exhaled breath analysis following metacholine challenge
  Interventions: Other: Metacholine challenge

INTERVENTIONS:
Other: Metacholine challenge — Exhaled breath analysis following metacholine challenge

SUMMARY:
This study is aiming at evaluating whether the number and size of exhaled particles changes during the increase and decrease of bronchial constriction in subjects with mild intermittent asthma.

DETAILED DESCRIPTION:
Particle emission demonstrates high reproducibility within subjects while between-subject-variability is large. Methacholine challenge in subjects with mild intermittent asthma will provide data from repetitive measurements in the same subject with variable airflow obstruction.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, aged 18 to 65 years.
2. Physician diagnosis of mild intermittent allergic asthma (GINA I according to GINA guidelines9).
3. Normal lung function parameters at baseline (FEV1 > 80 % of predicted)
4. Non smoker or smokers with a history of less than 10 pack years with no smoking in the last 12 months.
5. Able and willing to give written informed consent
6. Women will be considered for inclusion if they are:

not pregnant, as confirmed by pregnancy test, and not nursing of non-child bearing potential (i.e. physiologically incapable of becoming pregnant, including any female who is pre-menarchial or post-menopausal, with documented proof of hysterectomy or tubal ligation, or meet clinical criteria for menopause and has been amenorrhoeic for more than 1 year prior to the screening visit) of childbearing potential and using a highly effective method of contraception during the entire study (vasectomized partner, sexual abstinence - the lifestyle of the female should be such that there is complete abstinence from intercourse from two weeks prior to the study until at least 72 hours after the end of the study -, implants, injectables, combined oral contraceptives, hormonal IUDs, or double-barrier methods, i.e. any double combination of IUD, condom with spermicidal gel, diaphragm, sponge, and cervical cap)

• Available to complete all study measurements

Exclusion Criteria:

1. History of lower respiratory tract infection four weeks prior to the informed consent visit.
2. Past or present disease, which as judged by the investigator, may affect the outcome of this study. These diseases include, but are not limited to, cardiovascular disease, malignancy, hepatic disease, renal disease, hematological disease, neurological disease, endocrine disease or pulmonary disease (including but not confined to chronic bronchitis, emphysema, tuberculosis, bronchiectasis or cystic fibrosis).
3. Regular intake of any prescribed or over the counter medication. Exceptions include paracetamol for pain relief, oral contraceptive medication, hormonal replacement therapy, dietary and vitamin supplements, and short acting beta mimetics (SABA) on as needed basis.
4. Use of anti-inflammatory medication including systemic or inhaled corticosteroid within the last four weeks.
5. Any history of life-threatening asthma, defined as an asthma episode that required intubation and/or was associated with hypercapnea, respiratory arrest or hypoxic seizures.
6. Conditions or factors, which would make the subject unlikely to be able to undergo methacholine challenge.
7. Conditions which provide a contraindication for methacholine challenge testing such as uncontrolled arterial hypertension, known aortic aneurysm, myocardial infarction or stroke within three months prior to study, current use of cholinesterase inhibitor medication.
8. Inability to perform acceptable-quality spirometry.
9. History of drug or alcohol abuse.
10. Participation in another clinical trial 30 days prior to enrolment.
11. Suspected inability to understand the protocol requirements, instructions and study-related restrictions, the nature, scope, and possible consequences of the study.
12. Risk of non-compliance with study procedures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2010-03; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Exhaled breath analysis | Within one day
  In ten subjects with mild intermittent allergic asthma particles in exhaled breath will be analyzed for their number and size in a time dependent manner before and after induction of bronchial obstruction by methacholine challenge.

REFERENCES:
- See also: Related Info — http://www.atemwegsforschung.de